CLINICAL TRIAL: NCT03124407
Title: A Randomized, Multi-Dose, Placebo-Controlled Pain Relief Study of 0.25% 920-CGS-200 in Subjects With Preexisting Knee Pain (for at Least 6 Months) Caused by Osteoarthritis (OA)
Brief Title: Osteoarthritis Knee Pain Relief Study of 0.25% 920-CGS-200
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Propella Therapeutics (Industry)
Collaborators: Palm Beach Research, Inc (Unknown)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VZU-00022
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Results first posted 2020-03-30 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Knee
Keywords: knee pain, capsaicin, topical, osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Active treatment compared to drug vehicle as placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study medications were number coded only and identical in physical characteristics. Randomization coding was held only at the manufacturing site until data base lock.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Once daily-Active (Active Comparator): 40 subjects receiving once daily application of complete drug product (contains 0.25% capsaicin) to the knee
  Interventions: Drug: Capsaicin Topical Solution
- Once daily-Vehicle (Placebo Comparator): 20 subjects receiving once daily application of drug product vehicle (i.e., with no capsaicin) to the knee
  Interventions: Other: Drug product vehicle
- Twice daily-Active (Active Comparator): 40 subjects receiving twice daily application of complete drug product (contains 0.25% capsaicin) to the knee
  Interventions: Drug: Capsaicin Topical Solution
- Twice daily-Vehicle (Placebo Comparator): 20 subjects receiving twice daily application of drug product vehicle (i.e., with no capsaicin) to the knee
  Interventions: Other: Drug product vehicle

INTERVENTIONS:
Drug: Capsaicin Topical Solution — Over-the-counter Tentative Final Monograph compliant product with 0.25% capsaicin
  Arms: Once daily-Active; Twice daily-Active
Other: Drug product vehicle — This is the vehicle for the active treatment drug product, but without capsaicin
  Arms: Once daily-Vehicle; Twice daily-Vehicle

SUMMARY:
This is a study of an over-the-counter, capsaicin-based (0.25%) topical analgesic for management of osteoarthritis knee pain meeting the US Food and Drug Administration's (FDAs) Tentative Final Monograph (TFM) guidance for "External Analgesic Drug Products For Over-the-Counter Human Use," published in the Federal Register on February 8, 1983 (final proposed 21 CFR 348). Subjects meeting the inclusion criteria and not meeting the exclusion criteria were randomized into one of four groups: once daily treatment with active product, once daily treatment with product vehicle (no capsaicin), twice daily treatment with active product, and twice daily treatment with product vehicle (no capsaicin), all for 7 consecutive days of treatment. The twice daily treatments were spaced approximately 12 hours apart. Osteoarthritis knee pain was assessed by the 100 mm visual analog scale. Osteoarthritis knee pain assessments were done each day for 28 days. Tolerability data were also collected.

DETAILED DESCRIPTION:
This is a study of a over-the-counter, capsaicin-based (0.25%) topical analgesic for management of osteoarthritis knee pain meeting the US Food and Drug Administration's (FDAs) Tentative Final Monograph (TFM) guidance for "External Analgesic Drug Products For Over-the-Counter Human Use," published in the Federal Register on February 8, 1983 (final proposed 21 CFR 348). Subjects meeting the inclusion criteria and not meeting the exclusion criteria were randomized into one of four groups: once daily treatment with active product, once daily treatment with product vehicle (no capsaicin), twice daily treatment with active product, and twice daily treatment with product vehicle (no capsaicin), all for 7 consecutive days of treatment. The twice daily treatments were spaced approximately 12 hours apart. Both knees received study drug treatment but only one knee per subject was assigned as the "study knee".

Osteoarthritis knee pain was assessed by the 100 mm visual analog scale and the response criterion was a 50% or greater reduction in osteoarthritis knee pain from baseline. Baseline was defined as the visual analog scale recorded not more than 30 minutes before the first study drug application (on Study Day 1). For subjects in the once daily (QD) groups the osteoarthritis knee pain assessments were at 12 hrs after the initial application (during Study Day 1) and 24 hours (Study Day 2) after the initial application and then once in the morning on Study Days 3 - 28. For subjects in the twice daily (BID) groups the osteoarthritis knee pain assessments were at 12 hrs after the initial application (during Study Day 1) and 24 hours(Study Day 2) after the initial application and then once in the morning and once 12 hours later on Study Days 3 - 28.

Tolerability data were also collected as reported burning-stinging pain, erythema and pruritus at the site of application.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has granted written informed consent.
2. Subject is at least 18 years of age.
3. Subject has knee pain with radiographic evidence of osteoarthritis in at least one knee (including an x-ray within the previous 2 years).
4. Subject's osteoarthritis knee pain has been present for ≥ 6 months.
5. Subject has osteoarthritis knee pain of ≥ 50 mm in one knee based on the visual analog scale at screening.
6. Subject has regularly used topical over-the-counter pain relief products or over-the-counter oral medication (acetaminophen or ibuprofen) to treat/manage pain from osteoarthritis in the previous 3 months.
7. Subject is in good general health and free of any disease state or physical condition which, in the investigator's opinion, exposes the subject to an unacceptable risk by study participation.
8. Subject is capable of understanding and complying with all instructions and study procedures, including the ability to accurately evaluate their symptoms.
9. Subject must be a male or non-pregnant female. If female, subject must be past childbearing age or otherwise must test negative for pregnancy. Males and females must agree to use effective birth control during the study or for at least 30 days after last dose of study investigational product, if unable to complete the study.

Exclusion Criteria:

1. Subject has spontaneously improving or rapidly deteriorating osteoarthritis or knee pain.
2. Subject has rheumatoid or psoriatic arthritis, or a form of arthritis inconsistent with a diagnosis of osteoarthritis.
3. Subject has used any topical steroids on or in the vicinity of the knees within 1 week prior to Screening, or has had a knee injection within 1 month prior to Screening.
4. Subject is currently taking prescription pain medication.
5. Subject has shaved their knees within 2 days of first day of treatment (Day 1).
6. Subject has used any capsaicin containing product on or in the vicinity of the knees within 2 weeks prior to first day of treatment (Day 1).
7. Subject has used any topically applied products (including emollient/moisturizer) on or in the vicinity of the knees within 2 weeks prior to first day of treatment (Day 1).
8. Subject has used topical therapy on the knees that, in the investigator's opinion, might affect the study evaluations of signs and/or symptoms.
9. Subject has broken or damaged skin on their knees, or an open wound near the knees.
10. Subject has a history of allergy/sensitivity to topical substances.
11. Subject is not able to understand the nature, importance, or consequences of the study.
12. Subject has a psychiatric disorder or has significant anxiety or depression that, in the investigator's opinion, could interfere with the subject's ability to accurately assess their pain, adhere to study instructions, or complete the study.
13. Subject has hypertension that is not adequately controlled (medication to treat hypertension is allowed), vascular disease, psychological disorder, or other condition that, in the investigator's opinion, contraindicate the use of medication.
14. Is obese with a Body Mass Index (BMI) of greater than 40 kg/m2.
15. Subject requires a surgical procedure in the immediate future.
16. Subject is pregnant or nursing.
17. Subject has been treated with an investigational drug, device, or therapy within 30 days prior to first day of treatment (Day 1).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan A Ryan, Ph.D., Study Director — Palm Beach Research, Inc
Locations (3):
- United States (3):
  - Research Center, Clearwater, Florida
  - Research Center, Tampa, Florida
  - Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

RESULTS

PARTICIPANT FLOW:
Groups:
- QD-Active: 40 subjects receiving once daily application of complete drug product (contains 0.25% capsaicin) to the knee
  Capsaicin Topical Solution: OTC Tentative Final Monograph (TFM) compliant product with 0.25% capsaicin
- QD-Vehicle: 20 subjects receiving once daily application of drug product vehicle (i.e.. with no capsaicin) to the knee
  Drug product vehicle: This is the vehicle for the active treatment drug product
- BID-Active: 40 subjects receiving twice daily application of complete drug product (contains 0.25% capsaicin) to the knee
  Capsaicin Topical Solution: OTC Tentative Final Monograph (TFM) compliant product with 0.25% capsaicin
- BID-Vehicle: 20 subjects receiving twice daily application of drug product vehicle (i.e.. with no capsaicin) to the knee
  Drug product vehicle: This is the vehicle for the active treatment drug product
Period: Overall Study
Arm/Group | QD-Active | QD-Vehicle | BID-Active | BID-Vehicle
Started | 40 | 20 | 40 | 20
Completed | 39 | 20 | 39 | 20
Not Completed | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Once Daily-Vehicle: 20 subjects receiving once daily application of drug product vehicle (i.e., with no capsaicin) to the knee
  Drug product vehicle: This is the vehicle for the active treatment drug product, but with no capsaicin
- Twice Daily-Vehicle: 20 subjects receiving twice daily application of drug product vehicle (i.e. ,with no capsaicin) to the knee
  Drug product vehicle: This is the vehicle for the active treatment drug product, but with no capsaicin
- Total: Total of all reporting groups
Arm/Group | Once Daily-Active | Once Daily-Vehicle | Twice Daily-Active | Twice Daily-Vehicle | Total
Number analyzed (Participants) | 40 | 20 | 40 | 20 | 120
Age, Continuous [Mean (Full Range); unit: years] | 58.0 [35 to 90] | 55.2 [38 to 75] | 56.7 [36 to 74] | 56.5 [35 to 72] | 56.6 [35 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 10 | 27 | 10 | 73
  Male | 14 | 10 | 13 | 10 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 8 | 15 | 7 | 46
  White | 24 | 11 | 25 | 11 | 71
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 40 | 20 | 40 | 20 | 120
BMI (kg/m2) [Mean (Full Range); unit: kg/m^2] | 29.6 [20 to 39] | 28.9 [23 to 39] | 30.5 [19 to 40] | 29 [19 to 39] | 29.5 [19 to 40]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 50% or Greater Pain Score Reduction From Baseline to 24 Hours After First Dose of Study Drug Treatment.
Description: To evaluate the percentage of subjects who experience ≥50% reduction in osteoarthritis knee pain in the target knee compared with baseline at 24 hours following the first study drug treatment. Subjects in the once daily application group recorded their knee pain in a diary twice: at 12 hrs (± 1 hr) after their initial application and then again within ≤30 minutes before their daily topical application which was to be applied at 24 hrs (± 1 hr) after their previous day's application on all subsequent study days. Subjects in the twice daily application group recorded their knee pain in a diary within ≤30 minutes before each application on all study days. Subjects used a 100mm visual analogue scale when assessing their knee pain.
Time Frame: Study Day 2
Population: The analysis population included all subjects who received at least one application of study drug and reported a pain score on Study Day 2.
Measure: Number; unit: percentage of subjects
Groups:
- Twice Daily-Vehicle: 20 subjects receiving twice daily application of drug product vehicle (i.e., with no capsaicin) to the knee
  Drug product vehicle: This is the vehicle for the active treatment drug product, but with no capsaicin
Arm/Group | Once Daily-Active | Once Daily-Vehicle | Twice Daily-Active | Twice Daily-Vehicle
Number analyzed (Participants) | 37 | 20 | 39 | 20
percentage of subjects | 27.03 | 20.0 | 23.08 | 20.0

2. Secondary Outcome: Percentage of Subjects With 50% or Greater Pain Score Reduction From Baseline to Day 8 Post Study Drug Treatment.
Description: To evaluate the percentage of subjects who experience ≥50% reduction in osteoarthritis knee pain in the target knee compared with baseline after a 7 day period. Subjects in the once daily application group recorded their knee pain in a diary twice: at 12 hrs (± 1 hr) after their initial application and then again within ≤30 minutes before their daily topical application which was to be applied at 24 hrs (± 1 hr) after their previous day's application on all subsequent study days. Subjects in the twice daily application group recorded their knee pain in a diary within ≤30 minutes before each application on all study days. Subjects used a 100mm visual analogue scale when assessing their knee pain.
Time Frame: Study Days 1-7
Population: The analysis population included all subjects who received at least one application of study drug and reported pain scores during Study Days 1-7.
Measure: Number; unit: percentage of subjects
Groups:
- Once Daily-Active: 40 subjects receiving once daily application of complete drug product (contains 0.25% capsaicin) to the knee
  Capsaicin Topical Solution: OTC Tentative Final Monograph (TFM) compliant product with 0.25% capsaicin
- Once Daily-Vehicle: 20 subjects receiving once daily application of drug product vehicle (i.e.. with no capsaicin) to the knee
  Drug product vehicle: This is the vehicle for the active treatment drug product, but without capsaicin
- Twice Daily-Active: 40 subjects receiving twice daily application of complete drug product (contains 0.25% capsaicin) to the knee
  Capsaicin Topical Solution: OTC Tentative Final Monograph (TFM) compliant product with 0.25% capsaicin
- Twice Daily-Vehicle: 20 subjects receiving twice daily application of drug product vehicle (i.e.. with no capsaicin) to the knee
  Drug product vehicle: This is the vehicle for the active treatment drug product, but without capsaicin
Arm/Group | Once Daily-Active | Once Daily-Vehicle | Twice Daily-Active | Twice Daily-Vehicle
Number analyzed (Participants) | 38 | 20 | 38 | 20
percentage of subjects | 42.11 | 25 | 47.37 | 40

3. Secondary Outcome: Percentage of Subjects With 50% or Greater Pain Score Reduction From Baseline to Day 28 Post Study Drug Treatment.
Description: To evaluate the percentage of subjects who experience ≥50% reduction in osteoarthritis knee pain in the target knee compared with baseline after 28 days. Subjects in the once daily application group recorded their knee pain in a diary twice: at 12 hrs (± 1 hr) after their initial application and then again within ≤30 minutes before their daily topical application which was to be applied at 24 hrs (± 1 hr) after their previous day's application on all subsequent study days. Subjects in the twice daily application group recorded their knee pain in a diary within ≤30 minutes before each application on all study days. Subjects used a 100mm visual analogue scale when assessing their knee pain.
Time Frame: Study Days 1-28
Population: The analysis population included all subjects who received at least one application of study drug and reported any pain scores during the study.
Measure: Number; unit: percentage of subjects
Arm/Group | Once Daily-Active | Once Daily-Vehicle | Twice Daily-Active | Twice Daily-Vehicle
Number analyzed (Participants) | 40 | 20 | 40 | 20
percentage of subjects | 53.85 | 26.32 | 57.89 | 47.37

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of study drug treatment (Day 1) to the end of treatment (Day 28).
Description: Definition of adverse events were consistent with clinicaltrials.gov definitions. Application site adverse events were specifically collected at pre-application of study drug (-30 min (± 5 min), and at 15 (± 5 min), 30 (± 5 min), 45 (± 5 min), and 60 minutes (± 5 min) and after leaving the clinic on each day at home at the same time (± 2 hours) for 7 days.
Arm/Group | QD-Active | QD-Vehicle | BID-Active | BID-Vehicle
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20 | 0/40 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20 | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 26/40 | 9/20 | 35/40 | 13/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QD-Active (N=40) | QD-Vehicle (N=20) | BID-Active (N=40) | BID-Vehicle (N=20)
Application site pruritus (General disorders) | 7 | 4 | 5 | 1
Application site erythema (General disorders) | 1 | 0 | 13 | 1
Application site pain (General disorders) | 26 | 6 | 34 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No disclosure of any of the data and results of this STUDY by way of publication or otherwise, shall be made by RESEARCH CENTER, or any third party, without the prior written consent of VIZURI.